CLINICAL TRIAL: NCT05465057
Title: "HIIT Med Kiloene" Investigating the Physical, Metabolic, and Psychosocial Effects of High-intensity Interval Training (HIIT) in Childhood Obesity
Brief Title: "HIIT Med Kiloene".
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Steno Diabetes Centre North Denmark (Other); Aalborg University (Other); Municipalities of Northern Jutland, Denmark (Unknown); TrygFonden, Denmark (Industry); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Charlotte Nørkjær Eggertsen, MD, MD, Ph.d. stud., Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20200035
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Childhood; High Intensity Interval Training
MeSH Terms: conditions — Pediatric Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT + lifestyle intervention (Active Comparator): Allocation of HIIT training in conjuction with lifestyle intervention (TCOCT protocol) through computerbased randomization proces.
  Interventions: Behavioral: High intensity interval training (HIIT) + lifestyle intervention (TCOCT); Behavioral: Lifestyle intervention (TCOCT)
- Lifestyle intervention (Active Comparator): Allocation of lifestyle intervention (TCOCT protocol) through computerbased randomization proces.
  Interventions: Behavioral: Lifestyle intervention (TCOCT)

INTERVENTIONS:
Behavioral: High intensity interval training (HIIT) + lifestyle intervention (TCOCT) — The participants randomized for HIIT will perform supervised training sessions three times a week for 3 months. All HIIT programs consist of activities that involve 4 x 4 min. intervals at 90-95% of HRmax.
  The lifestyle intervention (TCOCT) comprises a lifestyle intervention targeting all aspects of everyday life, incl. guidance on diet, physical activity, sleep, screen time, and social problems. The participant will be scheduled for follow up in the out-patient clinic or municipal obesity clinic by a trained pediatric nurse and dietician after 6-12 weeks.
  Arms: HIIT + lifestyle intervention
Behavioral: Lifestyle intervention (TCOCT) — The lifestyle intervention (TCOCT) comprises a lifestyle intervention targeting all aspects of everyday life, incl. guidance on diet, physical activity, sleep, screen time, and social problems. The participant will be scheduled for follow up in the out-patient clinic or municipal obesity clinic by a trained pediatric nurse and dietician after 6-12 weeks.

SUMMARY:
In Denmark, 15% of children are overweight and 5% obese. Obese children and adolescents have several metabolic complications, such as pre-diabetes, hypertension, dyslipidaemia, and excess fat deposition in liver, already at a young age. In addition, obese children suffer from psychological issues such as low quality of life and anxiety. These findings underline the need for effective treatment strategies to eliminate the development of obesity-related complications.

We will conduct a two-study project in order to investigate the effect of high-intensity interval training (HIIT) and lifestyle intervention in obese children and adolescents on several metabolic risk factors and psychological problems.

Study 1 is a randomized controlled study including 150 obese children and adolescents recruited from the municipal obesity clinics in Northern Jutland. Study 1 will examine the value of a group based HIIT intervention in the children's local environment and investigate the association between HIIT and psychosocial wellbeing.

Study 2 is a randomized controlled study including 60 severe obese children and adolescents recruited from Videnscenter for Børn og Unge med Overvægt (VIBUO) at Aalborg University Hospital. Study 2 investigates the effect of HIIT and lifestyle intervention on metabolic and cardiovascular risk factors.

In both studies, the children and adolescents are 9-16 years old and will be randomized to lifestyle guidance or a combination of HIIT and lifestyle guidance for 3 months, both followed by 9 months of lifestyle guidance only.

Our primary goal is to show the efficacy of HIIT and facilitate the establishment of permanent targeted training propositions for obese children and adolescents with local anchoring in the municipalities.

DETAILED DESCRIPTION:
Purpose:

We will conduct a two-study project in order to investigate the effect of High-intensity interval training (HIIT) and lifestyle intervention in obese children and adolescents on several metabolic risk factors and psychological problems. Moreover, we wish to facilitate the establishment of permanent targeted training propositions for children and adolescents with obesity with local anchoring in the municipalities. Hereby, enhance and maintain the engagement of an active lifestyle throughout adolescence.

Study 1 will examine the value of a group based HIIT intervention in the children's local environment in addition to a validated lifestyle intervention protocol and investigate the association between HIIT, physical activity and quality of life. Moreover, we wish to investigate the applicability and adherence of the HIIT program in a community-based setting.

Study 2 will investigate the effect of a combined HIIT and validated lifestyle intervention on ectopic fat deposition, insulin sensitivity, inflammation, and muscle microvascular function in children with severe obesity. This study will give us a better understanding of the interplay between important components of the pathophysiology of obesity-related complications and the possible positive effects of HIIT intervention.

Background:

Treatment of childhood obesity Through the past 30 years, several studies have been conducted with various types of lifestyle interventions focusing on dietary modifications, increased psychical activity and behavioral therapy. A Cochrane Review from 2019, showed a significantly better result by multidisciplinary family-based intervention, who combined all three elements.

In Denmark an approach in obesity treatment, developed at The Children's Obesity Clinic, Regional Hospital Holbæk is commonly used.This method described in The Children's Obesity Clinic´s Treatment (TCOCT) protocol has shown positive results in both obtaining and maintaining weight loss in children with obesity. The treatment comprises a lifestyle intervention targeting all aspects of everyday life, incl. guidance on diet, physical activity, sleep, screen time, and social problems. However, training intervention is currently not part of the standard obesity treatment program offered to the majority of children with obesity in Denmark. In fact, no prior Danish study has examined the effects of HIIT, in combination with lifestyle intervention, on physiological and mental health in a large cohort of children and adolescents with obesity.

High-intensity interval training. High-intensity interval training is defined as intermittent exercise periods with intensities reaching 90-95% of maximal heart rate. Several studies show that HIIT induces weight reduction, cardiovascular health and quality of life. Obese children and adolescents are often discouraged from participating in sports, because of previous bad experiences and defeats. Therefore, a specialized group-based training set-up, where the children do not feel stigmatized and are able to socialize with peers, are essential for success.

Our previous study (Nordlet) examining 160 obese children with the TCOCT protocol found a significant better attention rate at the municipal clinics than at the university hospital, especially in the group of children of low social status. Hence, by placing the intervention in the local community, we work to limit the health inequality that many obese children experiences and increase the engagement and attention rate.

Psychosocial consequences of obesity intervention. Childhood and adolescence play a highly important role in the development of a balanced mental health. Despite this, the psychosocial impact of obesity is often an overlooked keystone in evaluation of the effect of lifestyle intervention programs. Former research have shown that obese children and adolescents often suffers from low quality of life and depression, which emphasizes the need for intervention.

In order to address psychosocial health, children suffering from obesity undergo a Beck Youth Inventory test, Pediatric Quality of life (PedsQl) and WHO-5 index as part of their obesity treatment at our center. WHO-5 index is a simple questionnaire with 5 subjects on well-being. The PedsQl is a validated questionnaire that evaluates aspects of quality of life through 23 questions. The Beck Youth Inventories test is a thorough questionnaire covering psychiatric symptoms such as depression and self-concept and enables an effect evaluation within these areas. None of the mentioned tests has, to our knowledge, been used in large-scale follow-up studies with HIIT and lifestyle intervention.

Obesity and metabolism Juvenile obesity is known to lead to cardiovascular and metabolic diseases in adulthood, but already in childhood metabolic complications are evident. The pathological mechanisms are hypothesized to be a result of lipotoxicity -the "sick fat theory". The sick fat theory describes the human inherent capacity to deposit excess energy as triglycerides in the subcutaneous adipose tissue, and exceeding this capacity leads to adipocyte apoptosis and attracting pro-inflammatory immune cells. When the subcutaneous storage capacity is exceeded, adipose tissue accumulates in organs such as liver and muscles, resulting in insulin resistance and non-alcoholic fatty liver disease (NAFLD). Even though this theory is plausible, it has not yet been fully tested in obese children. Advances in MRI technology allows now for non-invasive quantification of fat deposited in organs and muscles. Hereby it becomes possible to investigate the accumulation of fat and the effects of intervention in this context. Our research group has experience in a novel technique, named liquid biopsies, to measure liver and muscle cell derived circulating extracellular vesicles (EV), providing indirect measures of fat deposition in liver and muscles. Through advanced analysis of blood samples and specialized MRI modalities, we want to investigate the complex association of several physiological and metabolic parameters on obesity-related complications, and evaluate the effect of HIIT and lifestyle intervention on these interactions.

HIIT Protocol:

In each municipality, we will establish 1-3 teams covering different geographical areas. The training teams will comprise 6-10 children and adolescents. By placing the training teams in the children's immediate environment, we hope to facilitate social networking and include children from families from all social layers.

The children randomized for HIIT will perform supervised training sessions three times a week. All HIIT programs consist of activities that involve 4 x 4 min. intervals at 90-95% of HRmax, with 3 min active recovery in between each interval. Trainers will be physiotherapy students or students from the institute of Health Science and Technology at Aalborg University. All trainers will receive instructions to tailor the training interventions to inspire to high intensity physical activities.

The Danish Health Authority and TCOCT recommends 60 minutes of physical activity per day, but several studies have shown that this goal is difficult to maintain. In order to investigate sedentary behavior and level of activity outside the training facility, the children will be ask to wear an accelerometer (Axivity, AX3, Newcastle, UK) for 7 days at baseline, and after 3 and 12 month.

Normal-weight control group:

A normal-weight age matched control group will be included in study 2. However, these children will not undergo training sessions, but only MRI-investigations and blood sampling at baseline. We have chosen this procedure, since the investigations applied in the current study is rather new. Thus, representative reference values for extracellular vesicles and the reactive hyperemia (evaluated by MR-BOLD) is lacking.

Work packages (WP):

The project will be divided into six WP's.

WP 1: Clinical examination, HIIT intervention. WP 1 serve as the basis for all other WPs in the project. The schedule for obtaining outcome measures is described under each WP. In addition to data recordings during all training sessions, time points of data acquisition will be at baseline, 3 months, and 12 months.

All obese children enrolled in the project (both study 1 and 2) will initially undergo a treatment protocol that resembles the TCOCT protocol.

At baseline, anthropometrics (height, weight, waist and hip circumference, BMI, BMI-SDS), blood pressure, and pubertal stage data will be collected.

Immediately after baseline measurements the children will be randomized to either HIIT + TCOCT or TCOCT alone by a computerized randomisation procedure.

WP 2: Psychosocial effects of HIIT All the enrolled children and their primary caregiver will be ask to complete the WHO-5 index, Pediatric Quality of life (PedsQl) and Beck Youth Inventories test.

All questionnaires will be performed at baseline, and after 3 and 12 months to evaluate the short- and long-term psychosocial effects of HIIT. All questionnaires will be evaluated at the end of the project after 12 months.

WP 3: Inflammation, oxidative stress and insulin sensitivity. The children in study 2 will meet at the Department of Pediatrics, Aalborg University Hospital, to a one-day admission, in order to conduct all investigations within the same day to avoid a time bias. The children will meet after an overnight fast.

Trained staff will collect blood samples, in order to investigate standard-blood sample analysis, including glucose, HbA1C, parameters for liver and thyroid function, pro-inflammatory biomarkers, and extracellular vesicles.

All measurements will be analyzed at Dept. of Biochemistry, Aalborg University Hospital.

WP 4: Ectopic fat deposition. WP 4 consists of MRI scans of the abdomen and lower body to investigate the degree of fat deposited in the organs and muscles. Experienced personal at The Department of Radiology, Aalborg University Hospital, will perform all MR investigations.

To investigate extracellular vesicles from liver, muscles and their expression of pathophysiological relevant membrane proteins (e.g. CD36), laboratory analysis will be performed by small-particle flow cytometry on a high-sensitive flow cytometer.

WP 5: Muscle- and endothelial function. In relation to the MR-scans in WP 4, the children will undergo an MR BOLD, where imaging methods and a blood pressure cuff on the lower leg is used to investigate the degree of reactive hyperemia in the microvasculature.

WP 6: Evaluation of the anchoring process:

After termination of the project we will evaluate the established HIIT programs through continous dialog and work shops with the participating municipals.

Perspectives:

We expect that HIIT in combination with the TCOCT protocol will have significant effect on the children's well-being and quality of life. Moreover, we expect that the children will experience a BMI reduction and lower levels of metabolic and cardiovascular risk factors of obesity.

One of our primary goals is to show the efficacy of HIIT and the applicability of HIIT in community-based settings. Hereby, we pinpoint the importance of incorporation of physical activity in the treatment of obesity.

The results from this study will provide a greater understanding for the underlying mechanisms of obesity-related complications in children and adolescents with obesity. In addition, our findings may prove valuable in daily clinical practice in order to further individualize childhood obesity treatment and improve both preventive and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 90th percentile for study 1 and BMI > 99th percentile for age and gender for study 2.
* Age 9-16 years

Exclusion Criteria:

* Mental illness in the child, that complicates attendance at activities.
* Physical limitations or illness that prevent the child from performing high intensity training, e.g. broken limbs, known heart or lung disease, severe asthma, diabetes or metabolic disease.
* If participant is not able to perform all 12 weeks of exercise for other reasons.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in BMI and BMI z-score from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+ lifestyle intervention (TCOCT) group or the lifestyle intervention (TCOCT) group. | Baseline, 3 month and 12 month
  Our primary objective is to compare the change in BMI and BMI z-scores from baseline and three and 12-month follow-up between children randomized to either the HIIT+TCOCT group or the TCOCT group. BMI will be measured by Weight (kg) / Height (m) 2.
  Different measurements have been used throughout in the literature to assess childhood obesity. In BMI z-scores, the variation of BMI according to age and gender is accounted for. The variability of BMI z-scores have been shown to fall with increasing obesity, so a given change in BMI will correlate to a smaller change in BMI z-scores. We therefore decided to investigate our data using both BMI and BMI z scores as the primary outcomes.

SECONDARY OUTCOMES:
Changes in biochemical variables from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+TCOCT group or the TCOCT group. | Baseline, 3 month and 12 month
  As secondary objective, the changes in biochemical variables measuring inflammation, insulin sensitivity, lipidemia, thyroid function and adipocytokines, from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+TCOCT group or the TCOCT group, will be evaluated.
  We hypothesize that the findings will be more substantiated in children with obesity undergoing HIIT and TCOCT compared to only TCOCT.
  The biochemical measurements obtained will be:
  C-Reactive Protein (mg/l) hemoglobin (mml/l) white blood cell count (10E9/l) Uric acid (mmol/l) Interleukin 6,8,10,15 (pg/l) Glucose (mmol/l) HbA1C (mmol/mol) Insulin (pmol/l) C-peptide (mg/l) TSH (miu/l) ALAT (U/l) ASAT (U/l) Basp (U/l) LDH (U/l) GGT (U/l) Cholesterol total (mmol/l) Cholesterol LDL (mmol/l) Cholesterol HDL (mmol/l) Triglyceride (mmol/l) Leptin (µg/ml) Adiponectin (µg/ml)
Changes in blood pressure from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+TCOCT group or the TCOCT group. | Baseline, 3 month and 12 month
  As secondary objective, the changes in blood pressure from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+TCOCT group or the TCOCT group, will be analysed. We hypothesize that the findings will be more substantiated in children with obesity undergoing HIIT and TCOCT compared to only TCOCT.
Changes in MRI fat accumulation variables from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+TCOCT group or the TCOCT group | Baseline, 3 month and 12 month
  Quantification of liver fat, subcutaneous fat and visceral fat is performed using magnetic resonance imaging in a 3 Tesla MRI scanner (GE Premier) at Aalborg University Hospital. The participants is positioned supine on the scanner bed with a 30-channel (AIRTM) coil placed over the abdomen and a 60-channel in-bed coil. Proton-density fat fraction (PDFF) images will be obtained using a multi-point Dixon sequence (IDEAL IQ, axial direction), slice thickness 2 mm; TE min full; TR 5.9 ms; FOV 44 cm; acquisition matrix (160x160) generating in-phase and out-of-phase images and reconstruction of fat-only and water-only images as well as of a PDFF map.
  The software quantifing the amount of fat as cm2 by multiplying the cross-sectional areas of the pixels containing fat in the slice of interest.
Changes in variables for psychological problems and quality of life from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+ lifestyle intervention (TCOCT) group or the lifestyle intervention (TCOCT) group. | Baseline, 3 month and 12 month
  Changes in variables for psychological problems and health-related quality of life (HRQOL) from baseline and 3 and 12-month follow-up between the HIIT+TCOCT group or the TCOCT group, will be evaluated.
  Three validated questionnaires; WHO-5, Pediatric Quality of Life (PedsQL) and Beck Youth Inventories (BYI), is used to evaluate these parameters.
  WHO-5 evaluates quality of life through 5 questions. PedsQL is available for three different age groups and contains a parental proxy report. The score for PedsQL contains 3 subscores; physical functioning, psychosocial score, and total score. The raw score is on a 0-100 scale, where a higher score indicates a better health related quality of life.
  BYI is developed for children aged 7-18 years and contains of five self-reported inventories: depression, anxiety, anger, disruptive behavior, and self-concept. A raw score and a T-score is calculated for each inventory and a score > 55 indicates a risk of having a psychological problem.
Changes in level of general physical activity from baseline and 3 and 12-month follow-up between children randomized to either the HIIT+ lifestyle intervention (TCOCT) group or the lifestyle intervention (TCOCT) group. | Baseline, 3 month and 12 month
  Changes in level of general physical activity from baseline and 3 and 12-month follow-up will be measured by accelerometers (Axivity, AX3, Newcastle, UK).
  We hypothesis that HIIT intervention leads to an increase in the general physical activity level immediately after HIIT intervention at 3 months, and that this will sustain at 12 months follow-up.

OTHER OUTCOMES:
Comparison of the levels of biological and MRI parameters between the groups of children with obesity and a normal weight age matched control group. | Baseline
  As explorative objectives, we want to compare the levels of our different parameters (especially parametres of inflammation, extracellular vesicles and measurements of fat accumulation from MRI) between the groups of obese children and a normal weight control group.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Hagstrøm, MD, PHD, Study Director — Department of pediatrics, University hospital of Aalborg, Denmark
Locations (1):
- Department of Pediatrics, University Hospital of Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eggertsen CN, Vestergaard ET, Simonsen MB, Warner TC, Frokjaer JB, Handberg A, Olesen LG, Grontved A, Olesen AV, Hagstrom S, Brond JC, Larsen RG. Adding High-Intensity Interval Training to a Multidisciplinary Lifestyle Intervention for Childhood Obesity: Secondary Analysis of a Randomized Controlled Trial to Examine the Effects on Physical Activity Behavior. Scand J Med Sci Sports. 2026 Jan;36(1):e70185. doi: 10.1111/sms.70185. PMID 41460768